CLINICAL TRIAL: NCT00005403
Title: Heart Disease and the Black Health Disadvantage
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4320; R03HL046120 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To utilize national population data sets prepared by the National Center for Health Statistics, to (1) examine the current Black disadvantage in cardiovascular (CV) health, (2) explore potential clinical and epidemiologic causes, (3) incorporate emerging knowledge of new risk factors and (4) compare trends in medical treatment and risk factors for the four sex-race groups.

DETAILED DESCRIPTION:
BACKGROUND:

The Black health disadvantage remains a pressing public health issue in the United States. According to the Department of Health and Human Services 'Black and Minority Health Report', 65,000 excess deaths occur each year among Blacks when compared to the mortality experience of whites. Cardiovascular diseases make by far the largest contribution to this loss of life, accounting for over 30 percent of the excess. Despite improvements in CV mortality for all four major sex-race groups during the 1970's, the trends in heart disease in the United States began to diverge. A 50 percent slowing of the decline in coronary mortality occurred among Blacks from 1978-1986, compared to whites, and the gap in life expectancy between the races has widened. As noted in the 'Report', despite the widespread recognition of the importance of the problem, our knowledge regarding the causes of these differentials in CV disease was inadequate. To address this problem, the Report recommended support for 'innovative uses of current data' and 'cross-comparisons from different data sets', emphasizing the unique contribution population-based studies can make to 'understanding the health status and needs of minority populations'. Given the deterioration of the Black health status relative to the majority population, these recommendations took on new urgency.

DESIGN NARRATIVE:

Several separate analyses were conducted of prevalence surveys, epidemiologic followup studies, hospitalization surveys and vital statistics. These separate analyses were subsequently combined into a comprehensive description of the clinical and epidemiologic determinants of the Black CV disadvantage, and its future trends.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-02; Study Completion 1993-01 (Actual)

REFERENCES:
- [Background] Liao Y, Cooper RS. Continued adverse trends in coronary heart disease mortality among blacks, 1980-91. Public Health Rep. 1995 Sep-Oct;110(5):572-9; discussion 570-2. PMID 7480611